CLINICAL TRIAL: NCT02598960
Title: A Phase 1/2a Dose Escalation and Cohort Expansion Study for Safety, Tolerability, and Efficacy of BMS-986156 Administered Alone and in Combination With Nivolumab (BMS-936558, Anti PD-1 Monoclonal Antibody) in Advanced Solid Tumors
Brief Title: An Investigational Immuno-therapy Study of Experimental Medication BMS-986156, Given by Itself or in Combination With Nivolumab in Patients With Solid Cancers or Cancers That Have Spread.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA009-002; 2015-002505-11 (EudraCT Number)
Record Dates: First submitted 2015-10-21; First posted 2015-11-06 (Estimated); Results first posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BMS-986156: Dose Escalation (Experimental)
  Interventions: Drug: BMS-986156
- BMS-986156 + nivolumab (nivo): Dose Escalation (Experimental)
  Interventions: Drug: BMS-986156; Drug: Nivolumab
- BMS-986156: Dose Expansion (Experimental)
  Interventions: Drug: BMS-986156
- BMS-986156 + nivolumab (nivo): Dose Expansion (Experimental)
  Interventions: Drug: BMS-986156; Drug: Nivolumab
- BMS986156 + Nivo: Cohort Expansion (Experimental)
  Interventions: Drug: BMS-986156; Drug: Nivolumab

INTERVENTIONS:
Drug: BMS-986156
Drug: Nivolumab
  Arms: BMS-986156 + nivolumab (nivo): Dose Escalation; BMS-986156 + nivolumab (nivo): Dose Expansion; BMS986156 + Nivo: Cohort Expansion

SUMMARY:
The purpose of this study is to evaluate the safety and tumor-shrinking ability of experimental medication BMS-986156, when given by itself or in combination with nivolumab in patients with solid cancers that are advanced or cancers that have spread.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* For Dose Escalation:

  * Subjects with any previously treated advanced (metastatic or refractory) solid tumor
* For Cohort Expansion:

  * Subjects must have a previously treated advanced solid tumor to be eligible
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Willing and able to provide pre-treatment and on-treatment fresh tumor biopsy
* Women of child-bearing potential and men must use an acceptable method of contraception during treatment and for 23 weeks after treatment for women and 31 weeks for men

Exclusion Criteria:

* Known central nervous system metastases or central nervous system as the only source of disease
* Other concomitant malignancies (with some exceptions per protocol)
* Active, known or suspected autoimmune disease
* Uncontrolled or significant cardiovascular disease
* History of active or chronic hepatitis (e.g. Hep B or C)
* Impaired liver or bone marrow function
* Major surgery less than 1 month before start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2015-10-14 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (26):
- United States (7):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - UCSD Moores Cancer Center, La Jolla, California
  - Emory University, Atlanta, Georgia
  - The Ohio State University, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - The West Clinic, P.C., Germantown, Tennessee
- Australia (4):
  - Liverpool Cancer Therapy Center, Liverpool, New South Wales
  - Local Institution, Westmead, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Linear Clinical Research Ltd, Nedlands, Western Australia
- Local Institution - 0012, Ghent, Belgium
- Canada (2):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Toronto, Ontario
- France (3):
  - Local Institution, Paris
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Vlllejuif
- Germany (3):
  - Local Institution, Bonn
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Würzburg
- Italy (2):
  - Local Institution - 0015, Milan, Lombardy
  - Local Institution - 0014, Milan
- Local Institution, Amsterdam, Netherlands
- Local Institution, Madrid, Spain
- Switzerland (2):
  - Cantonal Hospital St. Gallen, Sankt Gallen
  - Local Institution, Zurich

REFERENCES:
- [Derived] Wang R, Baxi V, Li Z, Locke D, Hedvat C, Sun Y, Walsh AM, Shao X, Basavanhally T, Greenawalt DM, Patah P, Novosiadly R. Pharmacodynamic activity of BMS-986156, a glucocorticoid-induced TNF receptor-related protein agonist, alone or in combination with nivolumab in patients with advanced solid tumors. ESMO Open. 2023 Apr;8(2):100784. doi: 10.1016/j.esmoop.2023.100784. Epub 2023 Feb 28. PMID 36863094
- [Derived] Heinhuis KM, Carlino M, Joerger M, Di Nicola M, Meniawy T, Rottey S, Moreno V, Gazzah A, Delord JP, Paz-Ares L, Britschgi C, Schilder RJ, O'Byrne K, Curigliano G, Romano E, Patah P, Wang R, Liu Y, Bajaj G, Siu LL. Safety, Tolerability, and Potential Clinical Activity of a Glucocorticoid-Induced TNF Receptor-Related Protein Agonist Alone or in Combination With Nivolumab for Patients With Advanced Solid Tumors: A Phase 1/2a Dose-Escalation and Cohort-Expansion Clinical Trial. JAMA Oncol. 2020 Jan 1;6(1):100-107. doi: 10.1001/jamaoncol.2019.3848. PMID 31697308
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: BMS-986156 10mg: BMS-986156 10mg Q2W
- Part A: BMS-986156 30mg: BMS-986156 30mg Q2W
- Part A: BMS-986156 100mg: BMS-986156 100mg Q2W
- Part A: BMS-986156 240mg; Part C: BMS-986156 240mg: BMS-986156 240mg Q2W
- Part A: BMS-986156 800mg; Part C: BMS-986156 800mg: BMS-986156 800mg Q2W
- Part B: BMS-986156 30mg + Nivo 240mg: BMS986156 30mg Q2W + Nivo 240mg Q2W
- Part B: BMS-986156 100mg + Nivo 240mg: BMS986156 100mg Q2W + Nivo 240mg Q2W
- Part B: BMS-986156 240mg + Nivo 240mg; Part D: BMS-986156 240mg + Nivo 240mg: BMS986156 240mg Q2W + Nivo 240mg Q2W
- Part B: BMS-986156 800mg + Nivo 240mg: BMS986156 800mg Q2W + Nivo 240mg Q2W
- Part E: BMS-986156 480mg + Nivo 480mg: BMS986156 480mg Q4W + Nivo 480mg Q4W
Period: Treatment Period
Arm/Group | Part A: BMS-986156 10mg | Part A: BMS-986156 30mg | Part A: BMS-986156 100mg | Part A: BMS-986156 240mg | Part A: BMS-986156 800mg | Part C: BMS-986156 240mg | Part C: BMS-986156 800mg | Part B: BMS-986156 30mg + Nivo 240mg | Part B: BMS-986156 100mg + Nivo 240mg | Part B: BMS-986156 240mg + Nivo 240mg | Part B: BMS-986156 800mg + Nivo 240mg | Part D: BMS-986156 240mg + Nivo 240mg | Part E: BMS-986156 480mg + Nivo 480mg
Started (= Starting Initial Treatment Period) | 4 | 6 | 4 | 6 | 9 | 3 | 2 | 3 | 9 | 14 | 11 | 188 | 33
Completed (= completing initial treatment period) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 3 | 23 | 7
Not Completed | 4 | 6 | 4 | 6 | 9 | 2 | 2 | 3 | 7 | 11 | 8 | 165 | 26
Not completed — Disease Progression | 4 | 4 | 4 | 6 | 8 | 2 | 2 | 3 | 7 | 9 | 7 | 143 | 23
Not completed — Study drug toxicity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Not completed — Adverse Event unrelated to study drug | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 11 | 2
Not completed — participant request to discontinue | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Not completed — participant withdrew consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — No longer meets study criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other Reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Participants Entering Follow Up Period
Arm/Group | Part A: BMS-986156 10mg | Part A: BMS-986156 30mg | Part A: BMS-986156 100mg | Part A: BMS-986156 240mg | Part A: BMS-986156 800mg | Part C: BMS-986156 240mg | Part C: BMS-986156 800mg | Part B: BMS-986156 30mg + Nivo 240mg | Part B: BMS-986156 100mg + Nivo 240mg | Part B: BMS-986156 240mg + Nivo 240mg | Part B: BMS-986156 800mg + Nivo 240mg | Part D: BMS-986156 240mg + Nivo 240mg | Part E: BMS-986156 480mg + Nivo 480mg
Started (= participants entering follow up period) | 4 | 6 | 4 | 6 | 9 | 3 | 2 | 3 | 9 | 14 | 11 | 188 | 33
Completed | 3 | 6 | 4 | 6 | 9 | 3 | 2 | 3 | 9 | 13 | 10 | 159 | 28
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 29 | 5
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 11 | 2
Not completed — participant withdrew consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0
Not completed — lost to follow up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — follow up no longer required per protocol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Other Reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: BMS-986156 10mg | Part A: BMS-986156 30mg | Part A: BMS-986156 100mg | Part A: BMS-986156 240mg | Part A: BMS-986156 800mg | Part C: BMS-986156 240mg | Part C: BMS-986156 800mg | Part B: BMS-986156 30mg + Nivo 240mg | Part B: BMS-986156 100mg + Nivo 240mg | Part B: BMS-986156 240mg + Nivo 240mg | Part B: BMS-986156 800mg + Nivo 240mg | Part D: BMS-986156 240mg + Nivo 240mg | Part E: BMS-986156 480mg + Nivo 480mg | Total
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 9 | 3 | 2 | 3 | 9 | 14 | 11 | 188 | 33 | 292
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (18.57) | 59.7 (5.82) | 57.5 (10.08) | 49.5 (13.28) | 51.0 (13.82) | 58.3 (19.43) | 56.5 (9.19) | 50.7 (20.50) | 57.2 (12.09) | 55.6 (18.67) | 57.0 (9.30) | 59.0 (11.58) | 57.2 (13.05) | 57.9 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 1 | 3 | 5 | 1 | 1 | 2 | 4 | 5 | 7 | 100 | 22 | 156
  Male | 0 | 5 | 3 | 3 | 4 | 2 | 1 | 1 | 5 | 9 | 4 | 88 | 11 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
  Not Hispanic or Latino | 4 | 6 | 1 | 3 | 5 | 1 | 0 | 2 | 6 | 7 | 4 | 51 | 11 | 101
  Unknown or Not Reported | 0 | 0 | 1 | 3 | 4 | 2 | 2 | 1 | 3 | 7 | 7 | 136 | 21 | 187
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 13 | 5 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
  White | 3 | 6 | 3 | 5 | 8 | 3 | 2 | 3 | 8 | 12 | 11 | 171 | 27 | 262
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All Cause Adverse Events (AEs), Serious Adverse Events, AEs Leading to Discontinuation and Deaths
Description: Number of participants with all cause adverse events (AEs), serious adverse events (SAEs), adverse events leading to discontinuation, and number of participant deaths.
  AEs and laboratory values will be graded according to the NCI CTCAE version 4.03.
Time Frame: From first treatment to 100 days post last dose. Approximately 29 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: BMS-986156 10mg | Part A: BMS-986156 30mg | Part A: BMS-986156 100mg | Part A: BMS-986156 240mg | Part A: BMS-986156 800mg | Part C: BMS-986156 240mg | Part C: BMS-986156 800mg | Part B: BMS-986156 30mg + Nivo 240mg | Part B: BMS-986156 100mg + Nivo 240mg | Part B: BMS-986156 240mg + Nivo 240mg | Part B: BMS-986156 800mg + Nivo 240mg | Part D: BMS-986156 240mg + Nivo 240mg | Part E: BMS-986156 480mg + Nivo 480mg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 9 | 3 | 2 | 3 | 9 | 14 | 11 | 188 | 33
Participants
  Adverse Events (AEs) | 4 | 6 | 4 | 6 | 9 | 3 | 2 | 3 | 9 | 14 | 11 | 188 | 33
  Serious Adverse Events (SAEs) | 3 | 3 | 1 | 5 | 4 | 2 | 2 | 2 | 5 | 10 | 6 | 121 | 22
  AEs leading to Discontinuation | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 32 | 5
  Deaths | 4 | 5 | 3 | 5 | 6 | 2 | 2 | 3 | 6 | 11 | 8 | 141 | 27

2. Primary Outcome: Number of Participants With Laboratory Abnormalities in Specific Thyroid Tests
Description: Number of Participants with laboratory abnormalities in specific thyroid tests.
  TSH = Thyroid stimulating hormone ULN = Upper limit number LLN = Lower limit number
Time Frame: From first treatment to 100 days post last dose. Approximately 29 months
Population: All treated participants with at least one on - treatment TSH measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: BMS-986156 10mg | Part A: BMS-986156 30mg | Part A: BMS-986156 100mg | Part A: BMS-986156 240mg | Part A: BMS-986156 800mg | Part C: BMS-986156 240mg | Part C: BMS-986156 800mg | Part B: BMS-986156 30mg + Nivo 240mg | Part B: BMS-986156 100mg + Nivo 240mg | Part B: BMS-986156 240mg + Nivo 240mg | Part B: BMS-986156 800mg + Nivo 240mg | Part D: BMS-986156 240mg + Nivo 240mg | Part E: BMS-986156 480mg + Nivo 480mg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 9 | 3 | 2 | 3 | 9 | 14 | 11 | 188 | 33
Participants
  TSH > ULN | 1 | 2 | 0 | 2 | 2 | 0 | 0 | 1 | 1 | 4 | 5 | 72 | 19
  TSH > ULN WITH TSH ≤ ULN AT BASELINE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 42 | 11
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 37 | 9
  TSH < LLN | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 38 | 10
  TSH <LLN WITH TSH ≥ LLN AT BASELINE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 26 | 8
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 24 | 5

3. Primary Outcome: Number of Participants With Laboratory Abnormalities in Specific Liver Tests
Description: Number of Participants with laboratory abnormalities in specific liver tests.
  ALT = alanine aminotransferase AST = aspartate aminotransferase ALP = alkaline phosphatase
Time Frame: From first treatment to 100 days post last dose. Approximately 29 months
Population: All treated participants with at least one on - treatment liver test measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: BMS-986156 10mg | Part A: BMS-986156 30mg | Part A: BMS-986156 100mg | Part A: BMS-986156 240mg | Part A: BMS-986156 800mg | Part C: BMS-986156 240mg | Part C: BMS-986156 800mg | Part B: BMS-986156 30mg + Nivo 240mg | Part B: BMS-986156 100mg + Nivo 240mg | Part B: BMS-986156 240mg + Nivo 240mg | Part B: BMS-986156 800mg + Nivo 240mg | Part D: BMS-986156 240mg + Nivo 240mg | Part E: BMS-986156 480mg + Nivo 480mg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 9 | 3 | 2 | 3 | 9 | 13 | 11 | 188 | 33
Participants
  ALT OR AST > 3*ULN | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 25 | 3
  ALT OR AST> 5*ULN | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 2 | 14 | 1
  ALT OR AST> 10*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 6 | 0
  ALT OR AST > 20*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  TOTAL BILIRUBIN > 2*ULN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 5 | 1
  ALP > 1.5*ULN | 1 | 2 | 1 | 2 | 2 | 1 | 1 | 2 | 2 | 7 | 3 | 70 | 11
  ALT/AST ELEV>3*ULN;TOTAL BILIRUBIN>2*ULN IN 1 DAY | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 1
  ALT/AST ELEV>3*ULN;TOTAL BILIRUBIN>2*ULN IN 30 DAYS | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 1

4. Secondary Outcome: Best Overall Response
Description: BOR will be defined by CR, PR, PD and SD
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: From first dose to a response or progressive disease (Approximately 50 Months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: BMS-986156 10mg | Part A: BMS-986156 30mg | Part A: BMS-986156 100mg | Part A: BMS-986156 240mg | Part A: BMS-986156 800mg | Part C: BMS-986156 240mg | Part C: BMS-986156 800mg | Part B: BMS-986156 30mg + Nivo 240mg | Part B: BMS-986156 100mg + Nivo 240mg | Part B: BMS-986156 240mg + Nivo 240mg | Part B: BMS-986156 800mg + Nivo 240mg | Part D: BMS-986156 240mg + Nivo 240mg | Part E: BMS-986156 480mg + Nivo 480mg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 9 | 3 | 2 | 3 | 9 | 14 | 11 | 188 | 33
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 17 | 1
  Stable Disease | 2 | 1 | 2 | 1 | 4 | 1 | 0 | 2 | 2 | 6 | 6 | 59 | 12
  Progressive Disease | 1 | 3 | 2 | 4 | 4 | 2 | 2 | 0 | 4 | 4 | 4 | 91 | 15
  Not Evaluable | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 16 | 3
  Not Available | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

5. Secondary Outcome: Overall Response Rate
Description: Defined as the percentage of all treated participants whose BOR is either a complete response(CR) or partial response(PR).
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose to CR and PR (Approximately 50 Months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: BMS-986156 10mg | Part A: BMS-986156 30mg | Part A: BMS-986156 100mg | Part A: BMS-986156 240mg | Part A: BMS-986156 800mg | Part C: BMS-986156 240mg | Part C: BMS-986156 800mg | Part B: BMS-986156 30mg + Nivo 240mg | Part B: BMS-986156 100mg + Nivo 240mg | Part B: BMS-986156 240mg + Nivo 240mg | Part B: BMS-986156 800mg + Nivo 240mg | Part D: BMS-986156 240mg + Nivo 240mg | Part E: BMS-986156 480mg + Nivo 480mg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 9 | 3 | 2 | 3 | 9 | 14 | 11 | 188 | 33
Percentage of participants | 0 [0.0 to 60.2] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2] | 0 [0.0 to 45.9] | 0 [0.0 to 33.6] | 0 [0.0 to 70.8] | 0 [0.0 to 84.2] | 0 [0.0 to 70.8] | 11.1 [0.3 to 48.2] | 21.4 [4.7 to 50.8] | 9.1 [0.2 to 41.3] | 11.2 [7.0 to 16.6] | 9.1 [1.9 to 24.3]

6. Secondary Outcome: Progression Free Survival (PFS)
Description: The time from the first dosing date to the date of first objectively documented disease progression or death due to any cause, whichever occurs first.
  Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From first dose to disease progression (Approximately 50 Months)
Population: All treated participants with evaluable PFS measures
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A: BMS-986156 10mg | Part A: BMS-986156 30mg | Part A: BMS-986156 100mg | Part A: BMS-986156 240mg | Part A: BMS-986156 800mg | Part C: BMS-986156 240mg | Part C: BMS-986156 800mg | Part B: BMS-986156 30mg + Nivo 240mg | Part B: BMS-986156 100mg + Nivo 240mg | Part B: BMS-986156 240mg + Nivo 240mg | Part B: BMS-986156 800mg + Nivo 240mg | Part D: BMS-986156 240mg + Nivo 240mg | Part E: BMS-986156 480mg + Nivo 480mg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 9 | 3 | 2 | 3 | 9 | 14 | 11 | 188 | 33
Months | 3.48 [1.64 to NA] — Insufficient number of events to calculate | 1.74 [1.45 to NA] — Insufficient number of events to calculate | 2.66 [1.64 to NA] — Insufficient number of events to calculate | 1.64 [1.58 to NA] — Insufficient number of events to calculate | 1.84 [1.64 to 3.48] | 1.64 [1.64 to NA] — Insufficient number of events to calculate | 1.71 [NA to NA] — Insufficient number of events to calculate | 1.81 [1.64 to NA] — Insufficient number of events to calculate | 1.64 [0.89 to 22.47] | 3.71 [1.64 to 8.97] | 3.52 [1.61 to NA] — Insufficient number of events to calculate | 1.91 [1.81 to 3.25] | 2.92 [1.77 to 3.52]

7. Secondary Outcome: Duration of Response
Description: All treated participants with a BOR of CR or PR, is defined as the time between the date of first response and the date of disease progression or death, whichever occurs first.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose to disease progression after a response (Approximately 50 Months)
Population: All treated participants with a CR or PR
Measure: Median (Full Range); unit: Months
Arm/Group | Part A: BMS-986156 10mg | Part A: BMS-986156 30mg | Part A: BMS-986156 100mg | Part A: BMS-986156 240mg | Part A: BMS-986156 800mg | Part C: BMS-986156 240mg | Part C: BMS-986156 800mg | Part B: BMS-986156 30mg + Nivo 240mg | Part B: BMS-986156 100mg + Nivo 240mg | Part B: BMS-986156 240mg + Nivo 240mg | Part B: BMS-986156 800mg + Nivo 240mg | Part D: BMS-986156 240mg + Nivo 240mg | Part E: BMS-986156 480mg + Nivo 480mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 20 | 3
Months |  |  |  |  |  |  |  |  | 20.70 [20.7 to 20.7] | 30.10 [7.4 to 31.3] | NA [31.0 to 31.0] — Insufficient number of events to calculate | NA [0 to 31.8] — Insufficient number of events to calculate | NA [21.0 to 22.4] — Insufficient number of events to calculate

8. Secondary Outcome: Number of Participants With Anti-Drug Antibody Response
Description: Number of participants with a positive Anti-Drug Antibody to BMS-986156 or nivolumab
Time Frame: At Cycle 3 Day 1; where each treatment cycle was 8 weeks
Population: All BMS-986156 or Nivolumab Treated participants with Baseline and at Least One Post-baseline Assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: BMS-986156 10mg | Part A: BMS-986156 30mg | Part A: BMS-986156 100mg | Part A: BMS-986156 240mg | Part A: BMS-986156 800mg | Part C: BMS-986156 240mg | Part C: BMS-986156 800mg | Part B: BMS-986156 30mg + Nivo 240mg | Part B: BMS-986156 100mg + Nivo 240mg | Part B: BMS-986156 240mg + Nivo 240mg | Part B: BMS-986156 800mg + Nivo 240mg | Part D: BMS-986156 240mg + Nivo 240mg | Part E: BMS-986156 480mg + Nivo 480mg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 9 | 3 | 2 | 3 | 9 | 14 | 11 | 188 | 33
Participants
  BMS-986156: number analyzed (Participants) | 4 | 4 | 4 | 5 | 9 | 3 | 2 | 3 | 8 | 12 | 11 | 181 | 33
  BMS-986156 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0
  Nivolumab: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 8 | 11 | 11 | 171 | 33
  Nivolumab | 0 |  |  |  |  |  |  | 0 | 0 | 4 | 1 | 32 | 2

ADVERSE EVENTS:
Time Frame: AEs/SAEs are collected from the first dose date until the last dose date + 100 days. (Approximately up to 29 months)
Groups:
- Part A: BMS-986156 30mg: Part A: BMS-986156 30mg Q2W
- Part A: BMS-986156 240mg: Part A: BMS-986156 240mg Q2W
- Part B: BMS-986156 30mg +Nivo 240mg: BMS-986156 30mg Q2W +Nivo 240mg Q2W
- Part B: BMS-986156 100mg +Nivo 240mg: BMS-986156 100mg Q2W +Nivo 240mg Q2W
- Part B: BMS-986156 240mg +Nivo 240mg; Part D: BMS-986156 240mg +Nivo 240mg: BMS-986156 240mg Q2W +Nivo 240mg Q2W
- Part B: BMS-986156 800mg +Nivo 240mg: BMS-986156 800mg Q2W +Nivo 240mg Q2W
- Part E: BMS-986156 480mg +Nivo 480mg: BMS-986156 480mg Q4W +Nivo 480mg Q4W
Arm/Group | Part A: BMS-986156 10mg | Part A: BMS-986156 30mg | Part A: BMS-986156 100mg | Part A: BMS-986156 240mg | Part A: BMS-986156 800mg | Part C: BMS-986156 240mg | Part C: BMS-986156 800mg | Part B: BMS-986156 30mg +Nivo 240mg | Part B: BMS-986156 100mg +Nivo 240mg | Part B: BMS-986156 240mg +Nivo 240mg | Part B: BMS-986156 800mg +Nivo 240mg | Part D: BMS-986156 240mg +Nivo 240mg | Part E: BMS-986156 480mg +Nivo 480mg
All-Cause Mortality (participants affected / at risk) | 4/4 | 5/6 | 3/4 | 5/6 | 6/9 | 2/3 | 2/2 | 3/3 | 6/9 | 11/14 | 8/11 | 141/188 | 27/33
Serious Adverse Events (participants affected / at risk) | 3/4 | 3/6 | 1/4 | 5/6 | 4/9 | 2/3 | 2/2 | 2/3 | 5/9 | 10/14 | 6/11 | 121/188 | 22/33
Other Adverse Events (participants affected / at risk) | 4/4 | 5/6 | 4/4 | 6/6 | 9/9 | 3/3 | 1/2 | 2/3 | 8/9 | 14/14 | 11/11 | 185/188 | 31/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: BMS-986156 10mg (N=4) | Part A: BMS-986156 30mg (N=6) | Part A: BMS-986156 100mg (N=4) | Part A: BMS-986156 240mg (N=6) | Part A: BMS-986156 800mg (N=9) | Part C: BMS-986156 240mg (N=3) | Part C: BMS-986156 800mg (N=2) | Part B: BMS-986156 30mg +Nivo 240mg (N=3) | Part B: BMS-986156 100mg +Nivo 240mg (N=9) | Part B: BMS-986156 240mg +Nivo 240mg (N=14) | Part B: BMS-986156 800mg +Nivo 240mg (N=11) | Part D: BMS-986156 240mg +Nivo 240mg (N=188) | Part E: BMS-986156 480mg +Nivo 480mg (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Endocarditis noninfective (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ectopic antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatobiliary infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Stoma obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stoma site extravasation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1 | 2 | 3 | 1 | 2 | 2 | 3 | 4 | 2 | 72 | 13
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Thalamus haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ureteric haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Urogenital fistula (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: BMS-986156 10mg (N=4) | Part A: BMS-986156 30mg (N=6) | Part A: BMS-986156 100mg (N=4) | Part A: BMS-986156 240mg (N=6) | Part A: BMS-986156 800mg (N=9) | Part C: BMS-986156 240mg (N=3) | Part C: BMS-986156 800mg (N=2) | Part B: BMS-986156 30mg +Nivo 240mg (N=3) | Part B: BMS-986156 100mg +Nivo 240mg (N=9) | Part B: BMS-986156 240mg +Nivo 240mg (N=14) | Part B: BMS-986156 800mg +Nivo 240mg (N=11) | Part D: BMS-986156 240mg +Nivo 240mg (N=188) | Part E: BMS-986156 480mg +Nivo 480mg (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 2 | 30 | 5
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 3
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Eye discharge (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Periorbital swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 10 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0 | 2 | 3 | 0 | 0 | 0 | 1 | 3 | 2 | 22 | 9
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 8 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 10 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 2 | 1 | 0 | 0 | 3 | 1 | 2 | 28 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 4 | 1 | 0 | 0 | 1 | 4 | 3 | 35 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 4 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 2
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 1 | 3 | 2 | 1 | 0 | 0 | 4 | 5 | 5 | 44 | 12
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 1 | 1 | 8 | 2 | 28 | 8
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 27 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
Chills (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 4 | 2 | 15 | 2
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 1 | 2 | 3 | 2 | 1 | 1 | 1 | 5 | 7 | 57 | 15
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 11 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 3 | 25 | 6
Pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 17 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 3 | 3 | 0 | 0 | 2 | 3 | 5 | 5 | 34 | 3
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 8 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 11 | 4
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 20 | 6
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 8 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 7 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 11 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 11 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 7 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 9 | 2
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 5 | 4 | 34 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 9 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 6 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 20 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 5 | 25 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 8 | 5
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 9 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 4 | 11 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 15 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 11 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 11 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 10 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 5 | 3 | 22 | 3
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 6 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 7 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 6 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 12 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Kidney congestion (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 5 | 1 | 31 | 7
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 2 | 29 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 3
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 21 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 15 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 2
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 6 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vascular compression (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT02598960/Prot_SAP_000.pdf